CLINICAL TRIAL: NCT06594055
Title: Periodic Use of Continuous Glucose Monitoring With Personalized Diet Interventions Using AI Camera Among Non-insulin Treated Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Principal Investigator, Sun Joon, Moon, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KBSMC 2022-04-043
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; non-insulin; continuous glucose monitoring; AI camera; periodic use
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring; Blood Glucose Self-Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Control (Active Comparator): The control group used self-monitoring blood glucose (SMBG) for two weeks with a manual food diary, followed by diet education. They then repeated SMBG with a food diary three months later, with a final follow-up at the 6-month mark.
  Interventions: Device: Self-monitoring blood glucose; Device: Food diary
- Treatment 1 (Experimental): Treatment 1 group used CGM (Freestyle Libre) for two weeks with an AI food camera, followed by diet education. They then repeated CGM for two weeks with an AI food camera three months later, with a final follow-up at the 6-month mark.
  Interventions: Device: Continuous Glucose Monitoring; Device: AI food camera
- Treatment 2 (Experimental): Treatment 2 group used CGM for two weeks with an AI food camera, followed by diet education, without a repeat three months later. They had a final follow-up at the 6-month mark.
  Interventions: Device: Continuous Glucose Monitoring; Device: AI food camera

INTERVENTIONS:
Device: Continuous Glucose Monitoring — Continuous glucose monitoring is a wearable device that continuously collects glucose data from interstitial fluid.
  Arms: Treatment 1; Treatment 2
Device: Self-monitoring blood glucose — The control group used self-monitoring blood glucose (SMBG) for two weeks with a manual food diary, followed by diet education. They then repeated SMBG with a food diary three months later, with a final follow-up at the 6-month mark.
  Arms: Control
Device: AI food camera — The AI food camera automatically detects the contents and nutritional information of foods.
  Arms: Treatment 1; Treatment 2
Device: Food diary — A food diary is a record in which the user manually writes down the consumed foods and their amounts.
  Arms: Control

SUMMARY:
The aim of this study is to evaluate the periodic use of continuous glucose monitoring (CGM) with an AI camera and following diet education among non-insulin-treated type 2 diabetes patients.

DETAILED DESCRIPTION:
The control group used self-monitoring blood glucose (SMBG) for two weeks with a manual food diary followed by diet education and repeated SMBG with a food diary three months later. Treatment 1 group used CGM (Freestyle Libre) for two weeks with an AI food camera followed by diet education, and repeated CGM for two weeks with an AI food camera three months later. Treatment 2 group used CGM for two weeks with an AI food camera followed by diet education without repeat three months later. Every group followed at 6 months for the final outcome. HbA1c at 6 months is the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients
2. HbA1c 6.5% - 10%
3. No medication changes in the past 3 months, and receiving treatment with lifestyle modification or oral antidiabetic drugs or GLP-1 receptor agonists
4. Ages 18 - 80 years old

Exclusion Criteria:

1. Insulin users
2. Those who have used steroids within the past 3 months or are expected to use them during the study period (excluding ointments)
3. Type 1 diabetes patients
4. Patients who have undergone pancreatic resection
5. Patients undergoing hemodialysis or peritoneal dialysis
6. Those requiring continuous MRI and CT scans
7. Those deemed by the researcher to have difficulty handling continuous glucose monitors and AI cameras
8. Those deemed unsuitable for participation in this clinical trial by the investigator, other than those mentioned above
9. Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c between baseline and the 6-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group. | 6 month follow-up

SECONDARY OUTCOMES:
Change in HbA1c between baseline and the 6-month mark, non-inferiority comparison between treatment group 1 and treatment group 2. | 6 month follow-up
Change in HbA1c between baseline and the 3-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group. | 3 month follow-up
Change in blood pressure between baseline and the 6-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group | 6 month follow-up
Change in lipid parameters between baseline and the 6-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group | 6 month follow-up
Change in body weight between baseline and the 6-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group | 6 month follow-up
Change in waist circumference between baseline and the 6-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group | 6 month follow-up
Glycemic metrics of blinded CGM once at 6-month mark in treatment 1 group compared to control group, and treatment 2 group compared to control group | 6 month follow-up
Change in patient satisfaction questionnaires between baseline and the 6-month mark, comparison between groups. | 6 month follow-up
  Diabetes management self-efficacy scale (DMSES), appraisal of diabetes scale (ADS), and the summary of diabetes self-care activities measure (SDSCA) were used. DMSES has a 0-10 score scale for each item, with higher scores indicating better outcomes. ADS has a 1-5 score scale where lower scores are better in the psychological impact of diabetes subscale, and higher scores are better in the sense of self-control subscale. SDSCA has a 0-7 score scale for each item, with higher scores indicating better outcomes in the Diet, Exercise, Glucose monitoring, and Foot care subscales, while lower scores are better in the smoking subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuksamsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No